CLINICAL TRIAL: NCT00410124
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Study to Compare the Safety and Efficacy of RAD001 Plus Best Supportive Care (BSC) Versus BSC Plus Placebo in Patients With Metastatic Carcinoma of the Kidney Which Has Progressed on VEGF Receptor Tyrosine Kinase Inhibitor
Brief Title: RAD001 Plus Best Supportive Care (BSC) Versus BSC Plus Placebo in Patients With Metastatic Carcinoma of the Kidney Which Has Progressed After Treatment With Sorafenib and/or Sunitinib
Acronym: RECORD-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRAD001C2240; 2006-002070-21 (EudraCT Number)
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2012-12

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: advanced kidney cancer; everolimus; kidney cancer; oral therapy
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- RAD001 +BSC (Experimental): The study drugs were self administered by the patients. Patients were instructed to take the study drug as specified in the protocol. Patients were instructed to take two tablets (5 mg each) by mouth every day. Tablets were to be taken one tablet after another with a glass of water, at the same time each day in a fasting state or with a light fat-free meal. If disease progression occurred, patients were unblinded and if they were receiving RAD001, they would discontinue the study. Otherwise, they would be given the option to continue in the extension open label phase of 2 tablets of RAD001 5mg by mouth every day.
  Interventions: Drug: RAD001
- Placebo (plus BSC) (Placebo Comparator): Patients received matching placebo of RAD001 tablets twice a day along with Best Supportive Care. With the documented disease progression, the investigator could unblind the patient. If unblinded patient was receiving placebo treatment, they were given the option to continue in the extension open label phase of 2 tablets of RAD001 5mg by mouth every day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RAD001 — The dose of RAD001 was 10 mg/day. Patients were instructed to take two tablets (5 mg each) by mouth every day.
  Other Names: Everolimus
  Arms: RAD001 +BSC
Drug: Placebo
  Arms: Placebo (plus BSC)

SUMMARY:
To assess whether daily treatment with RAD001 could slow the growth and spread of metastatic carcinoma of the kidney. The safety of RAD001 was also to be studied in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic carcinoma and with histological or cytological confirmation of clear cell RCC (tissue from the original diagnosis of renal cell cancer is acceptable).
* The date of progression on sunitinib and/or sorafenib must be within 6 months.
* Patients may have received one or both agents
* Prior therapy with cytokines (i.e., IL-2, Interferon) and/or VEGF-ligand inhibitors (i.e., bevacizumab) are permitted.
* Prior vaccine therapy in the adjuvant setting is permitted.
* Patients with at least one measurable lesion at baseline as per the Response evaluation criteria in solid tumors (RECIST) criteria, either on physical exam or as determined by Computer Tomography (CT) Scan or Magnetic Resonance Imaging (MRI).
* Patients with a Karnofsky Performance Status ≥70%.
* Adequate bone marrow, liver and renal function.
* Patients with a life expectancy ≥ 3 months.
* Women of childbearing potential must have had a negative serum or urine pregnancy test 48 hours prior to the administration of the first study treatment.
* Patients who give a written informed consent obtained according to local guidelines

Exclusion Criteria:

* Patients currently receiving chemotherapy, immunotherapy, or radio-therapy or who have received these within 4 weeks of study entry
* Patients who have previously received mTOR inhibitors.
* Patients with a known hypersensitivity to RAD001 or other rapamycins (sirolimus, temsirolimus) or to its excipients.
* Patients with untreated CNS metastases or who are neurologically unstable despite treatment of the CNS metastases. (Patients with treated CNS metastases, who are neurologically stable off of corticosteroids, are eligible to enter study).
* Patients receiving chronic treatment with corticosteroids or another immunosuppressive agent
* Patients with a known history of HIV seropositivity.
* Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except low dose coumadin)
* Patients who have any severe and/or uncontrolled medical conditions
* Patients who have a history of another primary malignancy ≤ 3 years, with the exception of non-melanoma skin cancer, and carcinoma in situ of uterine cervix
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes.
* Patients who are using other investigational agents or who had received investigational drugs ≤ 4 weeks prior to randomization
* Patients unwilling to or unable to comply with the protocol

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (90):
- United States (30):
  - Novartis Investigative Site, Fayetteville, Arkansas
  - Novartis Investigative Site, Duarte, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Ocoee, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Columbia, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Bedford, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Tyler, Texas
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Morgantown, West Virginia
- Australia (6):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Woodville, South Australia
  - Novartis Investigative Site, Heidelberg, Victoria
- Canada (6):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, Alberta
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (8):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (6):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt/M
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
- Italy (8):
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Japan (13):
  - Novartis Investigative Site, Akita, Akita
  - Novartis Investigative Site, Chiba, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Sunto-gun, Shizuoka
  - Novartis Investigative Site, Utsunomiya, Tochigi
  - Novartis Investigative Site, Tokushima, Tokushima
  - Novartis Investigative Site, Chuo-ku, Tokyo
- Netherlands (4):
  - Novartis Investigative Site, Utrecht, Netherlands
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Nijmegen
- Poland (4):
  - Novartis Investigative Site, Gdañsk
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Spain (5):
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Spain
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia

REFERENCES:
- [Derived] Stein A, Bellmunt J, Escudier B, Kim D, Stergiopoulos SG, Mietlowski W, Motzer RJ; RECORD-1 Trial Study Group. Survival prediction in everolimus-treated patients with metastatic renal cell carcinoma incorporating tumor burden response in the RECORD-1 trial. Eur Urol. 2013 Dec;64(6):994-1002. doi: 10.1016/j.eururo.2012.11.032. Epub 2012 Nov 21. PMID 23219086
- [Derived] Stein A, Wang W, Carter AA, Chiparus O, Hollaender N, Kim H, Motzer RJ, Sarr C. Dynamic tumor modeling of the dose-response relationship for everolimus in metastatic renal cell carcinoma using data from the phase 3 RECORD-1 trial. BMC Cancer. 2012 Jul 23;12:311. doi: 10.1186/1471-2407-12-311. PMID 22824201
- [Derived] Oudard S, Thiam R, Fournier LS, Medioni J, Lamuraglia M, Scotte F, Fabre E, Kim D, Kpamegan E, Panneerselvam A, Cuenod CA. Optimisation of the tumour response threshold in patients treated with everolimus for metastatic renal cell carcinoma: analysis of response and progression-free survival in the RECORD-1 study. Eur J Cancer. 2012 Jul;48(10):1512-8. doi: 10.1016/j.ejca.2012.01.027. Epub 2012 Feb 16. PMID 22342553
- [Derived] Porta C, Calvo E, Climent MA, Vaishampayan U, Osanto S, Ravaud A, Bracarda S, Hutson TE, Escudier B, Grunwald V, Kim D, Panneerselvam A, Anak O, Motzer RJ. Efficacy and safety of everolimus in elderly patients with metastatic renal cell carcinoma: an exploratory analysis of the outcomes of elderly patients in the RECORD-1 Trial. Eur Urol. 2012 Apr;61(4):826-33. doi: 10.1016/j.eururo.2011.12.057. Epub 2012 Jan 5. PMID 22297244
- [Derived] Calvo E, Escudier B, Motzer RJ, Oudard S, Hutson TE, Porta C, Bracarda S, Grunwald V, Thompson JA, Ravaud A, Kim D, Panneerselvam A, Anak O, Figlin RA. Everolimus in metastatic renal cell carcinoma: Subgroup analysis of patients with 1 or 2 previous vascular endothelial growth factor receptor-tyrosine kinase inhibitor therapies enrolled in the phase III RECORD-1 study. Eur J Cancer. 2012 Feb;48(3):333-9. doi: 10.1016/j.ejca.2011.11.027. Epub 2011 Dec 30. PMID 22209391
- [Derived] White DA, Camus P, Endo M, Escudier B, Calvo E, Akaza H, Uemura H, Kpamegan E, Kay A, Robson M, Ravaud A, Motzer RJ. Noninfectious pneumonitis after everolimus therapy for advanced renal cell carcinoma. Am J Respir Crit Care Med. 2010 Aug 1;182(3):396-403. doi: 10.1164/rccm.200911-1720OC. Epub 2010 Mar 1. PMID 20194812
- [Derived] Motzer RJ, Escudier B, Oudard S, Hutson TE, Porta C, Bracarda S, Grunwald V, Thompson JA, Figlin RA, Hollaender N, Urbanowitz G, Berg WJ, Kay A, Lebwohl D, Ravaud A; RECORD-1 Study Group. Efficacy of everolimus in advanced renal cell carcinoma: a double-blind, randomised, placebo-controlled phase III trial. Lancet. 2008 Aug 9;372(9637):449-56. doi: 10.1016/S0140-6736(08)61039-9. Epub 2008 Jul 22. PMID 18653228

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Core period was terminated due to early achievements of efficacy targets and patients who were receiving study drug and patients receiving placebo in double blind phase had option to continue into the extension phase to receive open label RAD001.
Groups:
- RAD001 +BSC: The study drugs were self administered by the patients. Patients were instructed to take the study drug as specified in the protocol. Patients were instructed to take two tablets (5 mg each) by mouth every day. Tablets were to be taken one tablet after another with a glass of water, at the same time each day in a fasting state or with a light fat-free meal. If disease progression occurred at data cutoff of 28Feb2008, patients were unblinded and if they were receiving RAD001, they would discontinue the study. Otherwise, they would be given the option to continue in the extension open label phase of 2 tablets of RAD001 5mg by mouth every day.
- Placebo + BSC / RAD001: Patients received matching placebo of RAD001 tablets twice a day along with Best Supportive Care. With the documented disease progression at data cutoff of 28Feb2008, the investigator could unblind the patient. If unblinded patient was receiving placebo treatment, they were given the option to continue in the extension open label phase of 2 tablets of RAD001 5mg by mouth every day.
Period: Core Phase Double Blind (15 Months)
Arm/Group | RAD001 +BSC | Placebo + BSC / RAD001
Started | 277 (Started indicates randomized (FAS) and treated) | 139
Ongoing | 13 | 4
Completed Double Blind Treatment | 62 | 2
Completed | 75 (Patients ongoing/completed double blind phase had option entering extension phase continuing RAD001.) | 6 (All patients ongoing/completed/not completed in core had option to enter extension taking RAD001.)
Not Completed | 202 | 133
Not completed — Adverse Event | 36 | 2
Not completed — Abnormal Laboratory Value | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 13 | 2
Not completed — Lost to Follow-up | 4 | 0
Not completed — Administrative Problems | 2 | 0
Not completed — Death | 7 | 4
Not completed — Disease Progression | 137 | 124
Period: Extension Phase - Open Label (45 Months)
Arm/Group | RAD001 +BSC | Placebo + BSC / RAD001
Started | 67 | 111 (Patients on placebo in core received RAD001 in extension phase.)
Completed | 0 | 0
Not Completed | 67 | 111
Not completed — Adverse Event | 7 | 19
Not completed — Abnormal Laboratory Values | 0 | 1
Not completed — Abnormal Test Procedures | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 2 | 10
Not completed — Disease Progression | 56 | 78
Not completed — Patient no longer required study drug | 1 | 0
Not completed — Final Primary Analysis | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo + BSC: Patients received matching placebo of RAD001 tablets twice a day along with Best Supportive Care. With the documented disease progression, the investigator could unblind the patient. If unblinded patient was receiving placebo treatment, they were given the option to continue in the extension open label phase of 2 tablets of RAD001 5mg by mouth every day.
- Total: Total of all reporting groups
Arm/Group | RAD001 +BSC | Placebo + BSC | Total
Number analyzed (Participants) | 277 | 139 | 416
Age, Customized [Number; unit: participants]
  <65 years | 165 | 98 | 263
  >=65 years | 112 | 41 | 153
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 33 | 94
  Male | 216 | 106 | 322

OUTCOME MEASURES:

1. Primary Outcome: Progressive Free Survival (PFS) in Patients Who Receive RAD001 Plus Best Supportive Care(BSC) Versus Patients Who Receive Matching Placebo Plus BSC
Description: Progression Free survival is defined as the time from randomization to the date of first documented disease progression or death from any cause. The primary statistical analysis of PFS was based on central radiological assessments using a one-sided stratified log-rank test. Radiological assessments: every 8 weeks (+/-1 week) during the first year and every 12 weeks (+/- 1 week) during the second year and thereafter and at the end of the study. Kaplan-Meier methodology was used to estimate the median PFS for each treatment group.
Time Frame: Time from randomization to dates of disease progression, death from any cause or last tumor assessment reported between date of first patient randomized until 28Feb2008 cut of date.
Population: Full Analysis Set was performed on the intent-to-treat population which consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Placebo + BSC: Patients received matching placebo of RAD001 tablets twice a day along with Best Supportive Care. With the documented disease progression at data cutoff of 28Feb2008, the investigator could unblind the patient. If unblinded patient was receiving placebo treatment, they were given the option to continue in the extension open label phase of 2 tablets of RAD001 5mg by mouth every day.
Arm/Group | RAD001 +BSC | Placebo + BSC
Number analyzed (Participants) | 277 | 139
Months | 4.90 [3.98 to 5.52] | 1.87 [1.84 to 1.94]

2. Secondary Outcome: Overall Survival (OS) Assessed by the Monthly Overall Survival Assessments
Description: Overall survival (OS) was defined as the time from date of randomization to date of death due to any cause. Kaplan-Meier methodology was used to estimate the median overall survival for each treatment group
Time Frame: Assessed every month up to 2 years after the last patient was randomized into the study from the date of randomization to the time of death. (Data cutoff was 15Nov2009)
Population: Full analysis set was performed on the intent-to-treat population which consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | RAD001 +BSC | Placebo + BSC
Number analyzed (Participants) | 277 | 139
Months | 13.57 [11.96 to 17.87] | 13.01 [10.09 to 16.66]

3. Secondary Outcome: Best Overall Response Rate in Patients Who Receive RAD001 Plus BSC Versus Matching Placebo Plus BSC
Description: The Best Overall Response rate (BOR) is defined as the percentage of patients having achieved confirmed Complete Response + Partial Response. Complete Response (CR) = at least two determinations of CR at least 4 weeks apart before progression. • Partial response (PR) = at least two determinations of PR or better at least 4 weeks apart before progression. Radiological assessments: every 8 weeks (+/-1 week) during the first year and every 12 weeks (+/- 1 week) during the second year and thereafter and at the end of the study.
Time Frame: Time from randomization to dates of disease progression, death from any cause or last tumor assessment reported, between date of first patient randomized until 28Feb2008 cutoff date
Population: Full analysis set was performed on the intent-to-treat population which consisted of all randomized patients.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | RAD001 +BSC | Placebo + BSC
Number analyzed (Participants) | 277 | 139
Percentage of Participants | 1.8 [0.6 to 4.2] | 0.0 [NA to NA] — Upper and lower limit cannot be measured.

4. Secondary Outcome: Duration of Response in Patients Who Receive RAD001 Plus BSC Versus Placebo Plus BSC
Description: Duration of overall response (CR or PR) applies only to patients whose Best Overall Response (BOR) was Complete Response (CR) or Partial Response (PR). The start date is the date of first documented response (CR or PR) and the end date is the date of event defined as the first documented progression or death. Radiological assessments: every 8 weeks (+/-1 week) during the first year and every 12 weeks (+/- 1 week) during the second year and thereafter and at the end of the study.
Time Frame: as for outcome 3
Population: Full Analysis Set was performed on the intent-to-treat population which consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001 +BSC | Placebo + BSC
Number analyzed (Participants) | 5 | 0
months | NA [NA to NA] — No duration of response result due to small number of responders. |

5. Secondary Outcome: Analysis of Time to Definitive Deterioration of the Global Health Status/QoL Scale(QL) Scores of the EORTC QLQ-30 Questionnaire by at Least 10 Percent Using Kaplan Meier Method, by Treatment.
Description: The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) contains 30 items. These include a global health status/QoL scale, five functional scales, three symptom scales, and six single items. Global health status / QoL scale (QL), consisting of 2 questions each scored from 1 (very poor) to 7 (excellent), and with possible scores ranging from 2 to 14. Higher score indicates better functioning. Definitive deterioration by at least 10% is defined as a decrease in score by at least 10% compared to baseline, with no increase above this threshold observed during the course of the study. A single measure reporting a decrease of at least 10% is considered definitive only if it is the last one available for the patient. Time to definitive deterioration is the number of days between the date of randomization and date of assessment at which definitive deterioration is seen.
Time Frame: Baseline and every 28 days under treatment and at discontinuation from RAD001" until 28Feb2008 cutoff date
Population: Full Analysis Set was performed on the intent-to-treat population which consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001 +BSC | Placebo + BSC
Number analyzed (Participants) | 277 | 139
months | 4.76 (3.71) [3.71 to 6.47] | 3.91 (23.486) [2.79 to NA] — Upper limit was beyond the timeframe of the analysis.

6. Secondary Outcome: Time to Definitive Deterioration of the FKS-DRS Risk Score by at Least 2 Score Units Using Kaplan-Meier Method, by Treatment.
Description: The Functional Assessment of Cancer Therapy - Kidney Symptom Index, Disease Related Symptoms (FKSI-DRS) is a set of items to assess symptoms experienced by patients with advanced kidney cancer. These symptoms include fatigue, pain, weight loss, dyspnea, cough, fever and hematuria. There were 4 response categories (1=Not at all, 2= A little, 3=Quite a bit, 4=Very much), sum of item responses can range from 0 to 36. "0"= severely symptomatic patient and the highest score is an asymptomatic patient. Definitive deterioration of the FKSI-DRS score was defined as a decrease by at least 2 units compared to baseline, with no later increase above this threshold observed during the study. A single measure reporting a decrease of at least 2 units was considered definitive only if it is the last one available for the patient. Time to definitive deterioration is the number of days between the date of randomization and the date of the assessment at which definitive deterioration is seen.
Time Frame: Baseline and every 28 days under treatment and at discontinuation from RAD001" until 28Feb2008 cutoff date
Population: Full Analysis Set was performed on the intent-to-treat population which consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001 +BSC | Placebo + BSC
Number analyzed (Participants) | 277 | 139
months | 4.76 [3.75 to 7.39] | 3.84 [2.04 to 4.57]

7. Secondary Outcome: Time to Definitive Deterioration of the Physical Functioning Scale (PF)Score of the EORTC QLQ-C30 Questionnaire by at Least 10 Percent Using Kaplan_Meier Method, by Treatment.
Description: The EORTC QLQ-C30 contains 30 items. These include five functional scales (physical, role, emotional, social and cognitive functioning), three symptom scales fatigue, pain, nausea, and vomiting), a global health status/QoL scale, and six single items (dyspnea, diarrhea, constipation, anorexia, insomnia and financial impact). Physical Functioning (PF) sub-scale, consisting of 5 questions each scored from 1 (not at all) to 4 (very much), and with possible values ranging from 5 to 20. Definitive deterioration by at least 10% is defined as a decrease in score by at least 10% compared to baseline, with no later increase above this threshold observed during the course of the study. A single measure reporting a decrease of at least 10% is considered definitive only if it is the last one available for the patient. Time to definitive deterioration is the number of days between the date of randomization and the date of the assessment at which definitive deterioration is seen.
Time Frame: Baseline and every 28 days under treatment and at discontinuation from RAD001" until 28Feb2008 cutoff date
Population: Full Analysis Set was performed on the intent-to-treat population which consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001 +BSC | Placebo + BSC
Number analyzed (Participants) | 277 | 139
months | 5.06 [3.78 to 7.39] | 4.57 [2.79 to NA] — Upper limit could not be calculated.

8. Secondary Outcome: Pharmacokinetics of RAD001:Peak Concentration in a Dosing Interval (C-max); Pre-dose Concentration at 24-h Time Point in Dosing Interval (C-min) and Average Concentration in a Dosing Interval =(C-avg)
Description: Blood samples will be collected by direct venipuncture during regularly scheduled visits according to the collection plan provided in the study protocol. C-avg= Area under curve (AUC) in a dosing interval from time-zero to time of the last quantifiable concentration (AUC0-tlast)/ time of the last quantifiable concentration in a dosing interval (tlast)
Time Frame: At pre-dose and post-dose: 1 hour, 2 hour, 5 hour, 24 hour of Cycle 1 Day1, Cycle 1 Day 15 and at pre-dose from Cycle 2(day1) and all subsequent treatment cycles up until data cut-off 28 Feb 2008.
Population: The pharmacokinetics population consists of all patients who have a pharmacokinetic assessment with a sufficient number of evaluable blood samples. The analsyis was limited to RAD001 + BSC arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Day 1: Pharmacokinetic Blood Sampling: Full pharmacokinetic profile assessments on Cycle 1, Day 1 (at pre-dose and at 1h, 2h, 5h, and 24h post-dose) were performed. Troughs were collected for all patients on Day 1 of each treatment Cycle from month 2 until discontinuation from the study drug.
- Day 15: Pharmacokinetic Blood Sampling: Full pharmacokinetic profile assessments on Cycle 1, Day 15 (at pre-dose and at 1h, 2h, 5h, and 24h post-dose) were performed.
Arm/Group | Day 1 | Day 15
Number analyzed (Participants) | 13 | 12
ng/mL
  C-max | 68.1 (29.8) | 76.7 (39.3)
  C-min | 7.9 (3.4) | 19.8 (12.3)
  C-avg | 19.0 (7.0) | 30.4 (10.9)

9. Secondary Outcome: Pharmacokinetics of RAD001: Time at Which C-Max Occurs (t-Max)
Description: Blood samples will be collected by direct venipuncture during regularly scheduled visits according to the collection plan provided in the study protocol.
Time Frame: At pre-dose and post-dose: 1 hour, 2 hour, 5 hour, 24 hour of Cycle 1 Day 1, Cycle 1 Day 15 and at pre-dose of From Cycle 2 (Day 1) and all subsequent treatment cycles until data cut-off 28Feb2008.
Population: as for outcome 8
Measure: Median (Full Range); unit: h
Arm/Group | Day 1 | Day 15
Number analyzed (Participants) | 13 | 12
h | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 5.0]

10. Secondary Outcome: Pharmacokinetics of RAD001: Area Under Curve (AUC) in a Dosing Interval From Time-zero to Time of the Last Quantifiable Concentration. (AUC 0-tlast)
Description: as for outcome 9
Time Frame: At pre-dose and post-dose: 1 hour, 2 hour, 5 hour, 24 hour of Cycle 1 Day 1, Cycle 1 Day 15 and at pre-dose from Cycle 2 (Day 1) and all subsequent treatment cycles until data cut-off 28Feb2008.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Day 1 | Day 15
Number analyzed (Participants) | 13 | 12
ng.h/mL | 455.0 (168.5) | 729.1 (262.7)

11. Secondary Outcome: Pharmacokinetics of RAD001: Time of the Last Quantifiable Concentration in a Dosing Interval - (Tlast)
Description: as for outcome 9
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Median (Full Range); unit: hour
Arm/Group | Day 1 | Day 15
Number analyzed (Participants) | 13 | 12
hour | 24.0 [24.0 to 24.0] | 24.0 [24.0 to 24.0]

12. Secondary Outcome: Pharmacokinetics of RAD001: Apparent Systemic Clearance From Blood Following Extravascular Administration (CL/F)
Description: Blood samples will be collected by direct venipuncture during regularly scheduled visits according to the collection plan provided in the study protocol.Apparent oral clearance of RAD001 (CL/F) was calculated using AUC in a dosing interval of 24 hours (AUC0-24hours) value on Day 15 as: CL/F = dose/ AUC0-τ
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Day 15
Number analyzed (Participants) | 12
L/hour | 15.4 (5.3)

13. Secondary Outcome: Pharmacokinetics of RAD001: Normalized to Body Surface Area (CL/F)
Description: as for outcome 9
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L/hour/m^2
Arm/Group | Day 15
Number analyzed (Participants) | 12
L/hour/m^2 | 7.5 (2.3)

ADVERSE EVENTS:
Description: The Safety population consists of all patients who received at least one dose of study drug and who had at least one valid post-baseline safety assessment. Patients were analyzed according to the treatment actually received.
Groups:
- Randomized to RAD001+ BSC ( Blinded + Open Label): The study drugs were self administered by the patients. Patients were instructed to take the study drug as specified in the protocol. Patients were instructed to take two tablets (5 mg each) by mouth every day. Tablets were to be taken one tablet after another with a glass of water, at the same time each day in a fasting state or with a light fat-free meal. If disease progression occurred at data cutoff of 28Feb2008, patients were unblinded and if they were receiving RAD001, they would discontinue the study. Otherwise, they would be given the option to continue in the extension open label phase of 2 tablets of RAD001 5mg by mouth every day.
- Randomized to Placebo + BSC (Open Label): With the documented disease progression at data cutoff of 28Feb2008, the investigator could unblind the patient. If unblinded patient was receiving placebo treatment, they were given the option to continue in the extension open label phase of 2 tablets of RAD001 5mg by mouth every day.
- Randomized to Placebo + BSC (Double Blind Only): Patients received matching placebo of RAD001 tablets twice a day along with Best Supportive Care.
Arm/Group | Randomized to RAD001+ BSC ( Blinded + Open Label) | Randomized to Placebo + BSC (Open Label) | Randomized to Placebo + BSC (Double Blind Only)
Serious Adverse Events (participants affected / at risk) | 135/274 | 60/111 | 17/26
Other Adverse Events (participants affected / at risk) | 261/274 | 106/111 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized to RAD001+ BSC ( Blinded + Open Label) (N=274) | Randomized to Placebo + BSC (Open Label) (N=111) | Randomized to Placebo + BSC (Double Blind Only) (N=26)
Anaemia (Blood and lymphatic system disorders) | 13 | 5 | 0
Bone marrow reticulin fibrosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal effusion (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 0
Tongue oedema (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0
Asthenia (General disorders) | 4 | 1 | 2
Chest discomfort (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 4 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 7 | 0 | 0
General physical health deterioration (General disorders) | 3 | 1 | 2
Generalised oedema (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 2 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 4 | 0 | 0
Oedema peripheral (General disorders) | 3 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Performance status decreased (General disorders) | 1 | 2 | 0
Pyrexia (General disorders) | 13 | 5 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Biloma (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 2 | 0
Cholestasis (Hepatobiliary disorders) | 2 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 2 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0
Enterococcal infection (Infections and infestations) | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Incision site infection (Infections and infestations) | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 2 | 0
Lung infection (Infections and infestations) | 4 | 0 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0
Pleural infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 10 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0
Septic shock (Infections and infestations) | 3 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Wound abscess (Infections and infestations) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Device dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stent occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bile duct pressure increased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood amylase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood chloride decreased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 4 | 1 | 0
Blood urea increased (Investigations) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Cell death (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 9 | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pleura carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Coma (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 2 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 2 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 5 | 4 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 3 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Ureteric dilatation (Renal and urinary disorders) | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 11 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 11 | 2 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Shock (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized to RAD001+ BSC ( Blinded + Open Label) (N=274) | Randomized to Placebo + BSC (Open Label) (N=111) | Randomized to Placebo + BSC (Double Blind Only) (N=26)
Anaemia (Blood and lymphatic system disorders) | 108 | 42 | 4
Lymphopenia (Blood and lymphatic system disorders) | 29 | 7 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 19 | 8 | 0
Ear pain (Ear and labyrinth disorders) | 3 | 6 | 0
Abdominal pain (Gastrointestinal disorders) | 31 | 10 | 1
Abdominal pain upper (Gastrointestinal disorders) | 20 | 6 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 26 | 13 | 0
Constipation (Gastrointestinal disorders) | 60 | 25 | 5
Diarrhoea (Gastrointestinal disorders) | 90 | 28 | 2
Dry mouth (Gastrointestinal disorders) | 22 | 5 | 4
Haemorrhoids (Gastrointestinal disorders) | 17 | 1 | 0
Nausea (Gastrointestinal disorders) | 78 | 27 | 5
Stomatitis (Gastrointestinal disorders) | 106 | 33 | 3
Vomiting (Gastrointestinal disorders) | 63 | 19 | 3
Asthenia (General disorders) | 96 | 31 | 9
Fatigue (General disorders) | 86 | 40 | 8
General physical health deterioration (General disorders) | 6 | 3 | 2
Mucosal inflammation (General disorders) | 53 | 26 | 0
Non-cardiac chest pain (General disorders) | 12 | 8 | 0
Oedema peripheral (General disorders) | 79 | 25 | 5
Pyrexia (General disorders) | 55 | 24 | 1
Bronchitis (Infections and infestations) | 17 | 6 | 1
Nasopharyngitis (Infections and infestations) | 20 | 8 | 1
Urinary tract infection (Infections and infestations) | 14 | 5 | 0
Blood alkaline phosphatase increased (Investigations) | 11 | 6 | 0
Blood creatinine increased (Investigations) | 29 | 3 | 0
Gamma-glutamyltransferase increased (Investigations) | 20 | 7 | 0
Weight decreased (Investigations) | 27 | 19 | 2
Decreased appetite (Metabolism and nutrition disorders) | 82 | 24 | 6
Dehydration (Metabolism and nutrition disorders) | 9 | 5 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 10 | 4 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 60 | 21 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 36 | 15 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 45 | 17 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 18 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 | 20 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 13 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 11 | 9 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 14 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 8 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 8 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 34 | 17 | 3
Dizziness (Nervous system disorders) | 19 | 3 | 3
Dysgeusia (Nervous system disorders) | 32 | 14 | 1
Headache (Nervous system disorders) | 53 | 14 | 2
Paraesthesia (Nervous system disorders) | 12 | 1 | 2
Anxiety (Psychiatric disorders) | 14 | 3 | 2
Insomnia (Psychiatric disorders) | 30 | 11 | 2
Dysuria (Renal and urinary disorders) | 5 | 6 | 0
Haematuria (Renal and urinary disorders) | 4 | 0 | 2
Nocturia (Renal and urinary disorders) | 10 | 8 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 96 | 30 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 59 | 28 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 17 | 8 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 51 | 12 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 6 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 | 8 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 18 | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 38 | 14 | 3
Erythema (Skin and subcutaneous tissue disorders) | 15 | 2 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 20 | 7 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 16 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 43 | 12 | 2
Rash (Skin and subcutaneous tissue disorders) | 83 | 29 | 1
Hypertension (Vascular disorders) | 14 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.

The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.